CLINICAL TRIAL: NCT01925118
Title: Phase II Study of Irradiated Donor Lymphocyte Infusion Plus High-dose Interleukin-2 in Patients With Metastatic Malignant Melanoma and Renal Cell Carcinoma
Brief Title: Irradiated Donor Lymphocyte Infusion Plus High-dose IL-2
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Ineffectiveness
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Dae Seog Heo, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-1305-6130491
Record Dates: First submitted 2013-08-14; First posted 2013-08-19 (Estimated); Last update posted 2016-04-26 (Estimated); Status verified 2016-04

CONDITIONS: Metastatic Malignant Melanoma and Renal Cell Carcinoma
MeSH Terms: conditions — Melanoma; Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- High-dose IL-2 (Experimental)
  Interventions: Biological: Irradiated donor lymphocyte infusion

INTERVENTIONS:
Biological: Irradiated donor lymphocyte infusion

SUMMARY:
Partially HLA-matched irradiated donor lymphcyte infusion alone resulted in 27% overall response rate (ORR) in advanced renal cell carcinoma without significant toxicities. In addition, high-dose interleukin-2 (IL-2)showed an ORR of 6-21% in metastatic melanoma or renal cell carcinoma with a durable response in patients who achieved complete remission. Therefore, irradiated donor lymphocyte infusion plus high-dose IL-2 might show a synergistic anti-tumor activity agaist relapsed or metastatic melanoma or renal cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed malignant melanoma or renal cell carcinoma
* At stage IV or relapse
* At least one prior chemotherapy including targeted agents
* At least one haploidential or partially matched-HLA donor
* ECOG performance status 0-1
* Age 18-75 years
* Measurable lesion
* Adequate bone marrow, liver, and renal functions

Exclusion Criteria:

* Chemotherapy within 4 weeks
* Stem cell transplantation
* Active CNS metastasis
* Hypersensitivity to IL-2

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2013-08; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
12-week modified immune-related response rate | 12-week

SECONDARY OUTCOMES:
6-week modified immune-related response rate | 6-week
Overall response rate based on RECIST v1.1 | 6/12-week
Progression-free survival | 6-month
Overall survival | 1-year
Immune-related adverse events | 12-week

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea